CLINICAL TRIAL: NCT01360775
Title: Intervention of Nutritional Education Addressed to Carers of Dependant Patients
Brief Title: Nutritional Education for Dependant Patients
Acronym: atdom_nut
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Victoria Arija, Jordi Gol i Gurina Foundation
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PI09/90340
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2009-10

CONDITIONS: Risk of Malnutrition
Keywords: Nutritional status; Dependent patients; Nutritional educational intervention; Caregivers; Clinical assay
MeSH Terms: interventions — Nutrition Assessment

ARMS (2):
- nutritional counseling (Experimental): Supervision and monitoring of nutritional status of patients in the home care program, after making nutritional advice
  Interventions: Behavioral: nutritional counseling
- Not nutritional counseling (No Intervention)

INTERVENTIONS:
Behavioral: nutritional counseling — Nutritional counseling to caregivers of dependant patients at nutritional risk, Who were participants in the Home Care program conducted by nurses
  Arms: nutritional counseling

SUMMARY:
Objective: To assess the effect of a nutritional educational intervention on the risk of malnutrition dependent patients aimed at the caregivers.

Material and methods:

Intervention study with control group, with 200 patients randomized selected, in a Home Care Program of 5 Primary Care Centers, malnourished and dependents, older than 65 years and with a caregiver.

Socioeconomic and cultural characteristics of the patient and the caregiver are collected. Mini Nutritional Assessment (MNA), food intake, anthropometric and serum parameters of nutritional status: albumin, prealbumin, transferrin, hemoglobin, lymphocyte count, iron, ferritin, are evaluates on 0- 6-12 months. Also evaluated dentures, basic activities of daily living (Barthel test), cognitive state (Pfeiffer test) status of mood (Yesavage test).

Prior to the intervention, the educational procedure and the design of educational material are standardized among nurses. The nurses make an initial session for caregivers and monitored the education at home monthly (4 visits) up to 6 months. NANDA (NORTH AMERICAN NURSING DIAGNOSIS ASSOCIATION) specific methodology of the Nursing profession is used. The investigators studied the effect of the intervention on the caregivers on the patient's nutritional status by the MNA test, diet, anthropometry and biochemical parameters.

Bivariate normal test statistics and multivariate models were created to adjust the effect of the intervention.

The program SPSS / PC was used.

ELIGIBILITY:
Inclusion Criteria:

* Be included in the program ATDOM,
* 65 years or more,
* have an MNA between 17 and 23.5 points,
* have a caregiver.

Exclusion Criteria:

* have a MNA outside the range of 17 to 23.5 points,
* conducting enteral feeding
* have severe dysphagia,
* have any serious illness that progresses to malnutrition,
* take vitamin supplements and / or dietary supplements.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | at 0, 6 and 12 moths
  Nutritional status by : Mini Nutritional Assessment questionnaire (MNA validated questionaire), diet (validated questionaire), anthropometric measurements (weight, height, body circumferences) and biochemicals parametres (Serum albumin and serum prealbumin by chemiluminescence; serum transferrin by immunoturbidimetric; hemoglobin and lymphocyte count by coulter, serum iron by colorimetric using ferrozine, and serum ferritin by radioimmunoassay.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Centers, Tarragona and Reus, Tarragona, Spain

REFERENCES:
- [Derived] Fernandez-Barres S, Garcia-Barco M, Basora J, Martinez T, Pedret R, Arija V; Project ATDOM-NUT group. The efficacy of a nutrition education intervention to prevent risk of malnutrition for dependent elderly patients receiving Home Care: A randomized controlled trial. Int J Nurs Stud. 2017 May;70:131-141. doi: 10.1016/j.ijnurstu.2017.02.020. Epub 2017 Feb 23. PMID 28273591
- [Derived] Arija V, Martin N, Canela T, Anguera C, Castelao AI, Garcia-Barco M, Garcia-Campo A, Gonzalez-Bravo AI, Lucena C, Martinez T, Fernandez-Barres S, Pedret R, Badia W, Basora J. Nutrition education intervention for dependent patients: protocol of a randomized controlled trial. BMC Public Health. 2012 May 24;12:373. doi: 10.1186/1471-2458-12-373. PMID 22625878